CLINICAL TRIAL: NCT05501145
Title: Clinical Features, Outcomes, and Therapeutics of Ppregnancy-related Aortic Dissection
Brief Title: Clinical Features, Outcomes, and Therapeutics of Pregnancy-Related Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Other Study IDs: 5A Plan VII
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Aortic Dissection; Pregnancy Related
MeSH Terms: conditions — Aortic Dissection | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cesarean section and aortic repair — The timing of aortic repair and delivery have to be determined based on the type of the dissection, the stage of pregnancy (the gestation age), and the status of the fetus, as well as the level of local neonatal service.

SUMMARY:
Aortic dissection in pregnancy represents a lethal risk to both the mother and fetus, it has yet to yield the optimal therapeutic strategy. The aim of this study was to characterize the clinical features and outcomes in women with pregnancy-related acute aortic dissection, and to suggest therapeutic guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Women who presented with aortic dissection during pregnancy or post partum ≤12 weeks.

Exclusion Criteria:

* Loss of surgical information.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: From February 1 2012 through June 30 2022 for identification women who presented with aortic dissection during pregnancy or post partum ≤12 weeks
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong-jia Zhang, MD, Study Chair — Beijing Anzhen Hospital
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Beijing
  - Department of Obstetrics and Gynecology, Guangdong Provincial People's Hospital, Guangzhou
  - Department of Cardiac Surgery, Affiliated Hospital of Qingdao University, Qingdao
  - Department of Obstetrics and Gynecology, Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu H, Yang L, Chen CY, Qian SC, Ma LY, Diao YF, Wu XY, Wu SY, Dong ZQ, Shao YF, Zhang HJ, Sun LZ, Zhu JM, Zhang JR, Li H. Management strategies and outcomes in pregnancy-related acute aortic dissection: a multicentre cohort study in China. Heart. 2024 Oct 28;110(22):1298-1306. doi: 10.1136/heartjnl-2024-324009. PMID 39266045